CLINICAL TRIAL: NCT00792129
Title: A Multi-Center Study to Evaluate MiLIF(R) Versus Open Posterior Unilateral Lumbar Interbody Fusion (TLIF)
Brief Title: MIS MiLIF Versus Open
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ATV-03-002; 2007-003
Record Dates: First submitted 2008-11-13; First posted 2008-11-17 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Low Back Pain; Leg Pain
Keywords: MIS; Minimally invasive; Atavi; Flex Posure; retractor; Patients with chronic low back and/or leg pain who are candidates for elective lumbar interbody fusion through a posterior unilateral approach,; for inclusion in the study.; If the patient meets all of the eligibility criteria,; they will be enrolled into the study and have either the MiLIF or open procedure depending on the surgeon they present to; (i.e., what group their surgeon agreed to participate in.)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Posterior unilateral interbody fusion using an open approach midline incision (TLIF)
  Interventions: Device: The Atavi System
- Experimental: MiLIF procedure with specialized Atavi instrumentation and minimally invasive visualization capabilities
  Interventions: Device: The Atavi System

INTERVENTIONS:
Device: The Atavi System — The primary device in the Atavi system is the Flex Posture retractor and accessories such as dilators and an Expander Instrument.
  The Atavi System includes instruments used to access the spine by dilation of the overlying tissues, as well as a retracting device that is used to maintain the access. Once the retractor is in place, the visualization components of the system may be used.
  Other Names: MIS; Minimally invasive; Atavi; Flex Posure; retractor

SUMMARY:
This study is being undertaken to compare the clinical outcomes of patients that have unilateral posterolateral lumbar interbody fusion using a traditional open approach versus the MiLIF procedure based on the MiCOR Precision Bone Allograft, specialized Atavi instrumentation, and minimally invasive visualization capabilities.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized cohort design clinical study to evaluate the clinical outcomes of patients that have a minimally invasive lumbar interbody fusion (MiLIF) through the Atavi system compared to traditional unilateral open lumbar interbody fusion through a midline incision. the study will involve up to approximately 12 investigational sites and enroll up to 126 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 75 years of age
* Patient is scheduled for an elective spinal lumbar interbody single level fusion
* Patient is a candidate for posterior unilateral lumbar fusion through a midline incision
* Indication for surgery and dominant symptom of chronic low back and/or leg pain
* Diagnosis of one or more of the following:

  * Primary symptomatic degenerative disc disease confirmed with appropriate imaging studies and/or positive lumbar discography
  * Spondylolisthesis Grade I/II
* The affected motion segment reside in L2-S1 and are adjacent segments
* Patient, or authorized representative, signs a written Informed Consent form to participate in the study, prior to any study mandated determinations or procedure.

Exclusion Criteria:

* Patient has a known fracture in the lumbar spine
* Patient has systemic infection or evidence of any surgical site infection (superficial or organ space)
* Patient has compromised immune system or autoimmune disease (WBC<4000 or >20,000)
* Patient has uncontrolled diabetes
* Patient has a known malignancy
* Prior lumbar fusion attempt; prior laminectomy and/or discectomy are allowed
* Known medical or anatomical condition that would preclude a posterior lumbar fusion using metallic instrumentation (e.g., severe osteopenia)
* Patient with a planned placement of an electric bone stimulator
* Patient with a planned placement of indwelling epidural catheter for a long term pain management
* Patient is pregnant or wishes to become pregnant during the length of the study participation
* Patient is currently in litigation
* Patient is not likely to comply with the follow-up evaluation schedule
* Patient is participating in a clinical trial of another investigational drug or device.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic low back and/or leg pain who are candiates for elective lumbar interbody fusion through a postierior unilateral approach, that present to either group of surgeons, will be screened for inclusion in the study. If the patient meets all of the eligibility criteria, they wil be enrolled into the study and have either the MiLIF or open procedure depending on the surgoen they present to (i.e., what group their surgeon agreed to participate in).
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2004-04; Primary Completion 2006-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Clinical Outcomes | MiLIF and Open groups at 3 months post-procedure as defined by the mean Oswestry score

SECONDARY OUTCOMES:
Clinical Outcomes | The percent of patients that have a successful fusion at one year post-procedure as measured by radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Joe Murar, M.D., Study Director — Zimmer Spine
Locations (9):
- United States (9):
  - La Jolla Spine Institute, La Jolla, California
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - Advanced Orthopedic Center, Port Charlotte, Florida
  - Southeastern Spine Center, Sarasota, Florida
  - Kennedy-White Orthopedic, Sarasota, Florida
  - Oregon Brain & Spinal Institute, Portland, Oregon
  - Williamette Neurosurgery, Salem, Oregon
  - William Beaumont Army Medical Center, El Paso, Texas
  - Naval Medical Center, Portsmouth, Virginia